CLINICAL TRIAL: NCT00945100
Title: Increasing Patching for Amblyopia in Children 3 to < 8 Years Old
Acronym: ATS15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-143; 2U10EY011751 (NIH)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; patching; occlusion
MeSH Terms: conditions — Amblyopia; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): 2 hours daily patching
  Interventions: Device: Eye Patch
- Intensified treatment (Active Comparator): 42 hours per week of patching (averaging 6 hours daily)
  Interventions: Device: Eye Patch

INTERVENTIONS:
Device: Eye Patch — 42 hours patching per week (averaging 6 hours patching daily)
  Other Names: Coverlet; 3M Opticlude; Ortopad
  Arms: Intensified treatment
Device: Eye Patch — 2 hours patching daily
  Other Names: Coverlet; 3M Opticlude; Ortopad
  Arms: Control

SUMMARY:
This study is designed to evaluate the effectiveness of increasing prescribed patching treatment from 2 to 6 daily hours after visual acuity has stabilized with initial treatment and amblyopia is still present. Children ages 3 to <8 years with visual acuity of 20/50 to 20/400 in the amblyopic eye will be enrolled in a run-in phase with 2 hours daily patching until no improvement, followed by randomization of eligible patients to patching 2 hours daily versus an average of 6 hours daily (42 hours per week). The primary objective is to determine if increasing patching dosage will improve visual acuity in patients with amblyopia still present after visual acuity has stabilized with initial treatment.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Both patching and atropine are accepted treatment modalities for the management of moderate amblyopia in children.1 Many practitioners prescribe 2 hours daily patching as initial therapy for amblyopia. However, many children fail to achieve normal visual acuity in the amblyopic eye with this regimen. In a randomized trial conducted by PEDIG comparing patching regimens, 71 of 92 patients with moderate amblyopia (77%) had amblyopic eye visual acuity of 20/32 or worse after 4 months of patching 2 hours daily.2 In another PEDIG randomized trial comparing patching to spectacles alone after a period of refractive adaptation, patients were treated with 2 hours daily patching and followed every 5 weeks until there was no improvement in amblyopic eye acuity. Fifty-five of 70 patients with moderate amblyopia (79%) and 14 of 14 patients with severe amblyopia (100%) had best-measured amblyopic eye visual acuity of 20/32 or worse after a median treatment period of 10 weeks.3 When improvement with initial therapy stops and amblyopia is still present, treatment options include increasing the dosage of current treatment, switching to another treatment, maintaining the same treatment and dosage for additional months, or combining treatments. Many clinicians will choose to increase the dosage of the current treatment, in part because families have become comfortable with that particular mode of treatment. However, it is unknown whether increasing occlusion dosage will improve amblyopic eye visual acuity in these patients. We are unaware of any reports of response to intensified treatment of amblyopia.

ELIGIBILITY:
Inclusion Criteria:

Major Eligibility Criteria for Run-in Phase

* Age 3 to < 8 years
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye between 20/50 and 20/400 inclusive
* Visual acuity in the sound eye 20/32 or better and inter-eye acuity difference >3 logMAR lines
* Amblyopia treatment within the past 6 months subject to the following stipulations:

  * No more than 6 weeks of any amblyopia treatment other than spectacles (except for patients being treated with 2 hours of patching per day who are entering the study on treatment)
  * No simultaneous treatment with patching and atropine
  * No use of atropine in combination with the sound eye spectacle lens reduced by more than 1.50 D
  * Maximum level of treatment within the past 6 months:

    * Patching: up to 2 hours daily
    * Atropine: up to once daily
* Wearing spectacles with optimal correction (if applicable); if amblyopic eye acuity is 20/80 or better, then VA must be stable in glasses. If amblyopic eye acuity is 20/100 or worse, then spectacles and patching can be initiated simultaneously.

Eligibility Criteria for Randomization:

* Amblyopic eye acuity of 20/40 to 20/160 with an inter-ocular difference of >2 lines, or amblyopic eye acuity of 20/32 with 3 lines of IOD.
* Reasonable compliance with prescribed treatment, defined as wearing the patch at least 10 hours per week.

Exclusion Criteria:

* Currently using vision therapy or orthoptics
* Ocular cause for reduced visual acuity (nystagmus per se does not exclude the patient if the above visual acuity criteria are met)
* Prior intraocular or refractive surgery
* Known skin reaction to patch or bandage adhesives

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K. Wallace, M.D., Study Chair — Duke University Eye Center
Locations (2):
- United States (2):
  - Southern California College of Optometry, Fullerton, California
  - Duke University Eye Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website at http://pedig.jaeb.org/Studies.aspx?RecID=29

REFERENCES:
- [Background] Wallace DK, Lazar EL, Crouch ER 3rd, Hoover DL, Kraker RT, Tamkins SM; Pediatric Eye Disease Investigator Group. Time course and predictors of amblyopia improvement with 2 hours of daily patching. JAMA Ophthalmol. 2015 May;133(5):606-9. doi: 10.1001/jamaophthalmol.2015.6. No abstract available. PMID 25695355
- [Result] Pediatric Eye Disease Investigator Group; Wallace DK, Lazar EL, Holmes JM, Repka MX, Cotter SA, Chen AM, Kraker RT, Beck RW, Clarke MP, Lorenzana IJ, Petersen DB, Roberts JT, Suh DW. A randomized trial of increasing patching for amblyopia. Ophthalmology. 2013 Nov;120(11):2270-7. doi: 10.1016/j.ophtha.2013.04.008. Epub 2013 Jun 4. PMID 23755872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2009 and December 2012, 45 sites randomized 169 participants to either increase patching time to an average of 6 hours per day (n=86) or continue 2 hours daily patching (n=83).
Pre-assignment Details: Prior to being considered for the randomized trial, participants who had not already completed at least 12 weeks of 2 hours of daily patching were enrolled into a run-in phase and treated with 2 hours of daily patching (and spectacles if needed) with follow-up every 6 weeks until no improvement.
Period: 10-week Primary Outcome
Arm/Group | Control | Intensified Treatment
Started | 83 | 86
Completed, Eligible | 55 (Eligible for Post-10 week phase) | 63 (Eligible for Post-10 week phase)
Completed, Not Eligible | 27 (Not Eligible for Post-10 week phase) | 20 (Not Eligible for Post-10 week phase)
Completed | 82 | 83
Not Completed | 1 | 3
Period: Post-10 Week Primary Outcome
Arm/Group | Control | Intensified Treatment
Started | 55 (27 participants were not eligible for Post 10 week Primary Outcome phase) | 63 (20 participants were not eligible for Post 10 week Primary Outcome phase)
Completed | 51 | 56
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intensified Treatment | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 83 | 86 | 169
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (1.3) | 5.9 (1.2) | 5.9 (1.3)
Age, Customized [Number; unit: participants] — Baseline age reflects age at randomization.
  The age eligibility requirement at enrollment was 3 to <8 years old, however, there were 7 participants who were enrolled into the run-in phase that were 8 years old by the time they were randomized.
  participants
    3 to <4 years | 5 | 8 | 13
    4 to <5 years | 15 | 15 | 30
    5 to <6 years | 27 | 19 | 46
    6 to <7 years | 17 | 25 | 42
    7 to 8 years | 19 | 19 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 40 | 43 | 83
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57 | 66 | 123
  Black/African American | 8 | 2 | 10
  Hispanic | 14 | 14 | 28
  Asian | 2 | 3 | 5
  More than one race | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 80 | 82 | 162
  United Kingdom | 3 | 3 | 6
  Canada | 0 | 1 | 1
Enrollment Disposition [Number; unit: participants] — Participants were classified into 3 groups (no current treatment, on treatment, ready for randomization) according to their treatment disposition at enrollment.
  participants
    No current treatment | 48 | 49 | 97
    On treatment | 18 | 18 | 36
    Ready for randomization | 17 | 19 | 36
Duration of patching prior to randomization (weeks) [Number; unit: participants]
  12 to <16 weeks | 14 | 21 | 35
  16 to <25 weeks | 39 | 31 | 70
  25 weeks or more | 30 | 34 | 64
Duration of patching prior to randomization (weeks) [Mean (Standard Deviation); unit: Weeks] | 24.5 (10.7) | 24.4 (11.9) | 24.4 (11.3)
Amblyopia Cause [Number; unit: participants] — Amblyopia associated with strabismus (comitant or incomitant), anisometropia, or both:
  Criteria for strabismus: At least one of the following:
  1. Heterotropia at distance and/or near fixation on examination (with or without spectacles)
  2. History of strabismus surgery
  3. Documented history which is no longer present (which in the judgement of the investigator could have caused amblyopia)
  Criteria for anisometropia: At least one of the following:
  1. At least 0.50 D difference between eyes in spherical equivalent
  2. At least 1.50 D different between eyes in astigmatism in any meridian
  participants
    Strabismus | 16 | 16 | 32
    Anisometropia | 41 | 34 | 75
    Strabismus and Anisometropia | 26 | 36 | 62
Best distance visual acuity in the amblyopic eye at randomization [Number; unit: participants] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction (if applicable) by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  Best amblyopic eye visual acuity was computed as the better of the initial test and retest visual acuities at randomization.
  participants
    20/160 | 2 | 3 | 5
    20/125 | 3 | 1 | 4
    20/100 | 2 | 7 | 9
    20/80 | 6 | 6 | 12
    20/63 | 17 | 21 | 38
    20/50 | 26 | 24 | 50
    20/40 | 21 | 18 | 39
    20/32 | 6 | 6 | 12
Best distance visual acuity in the amblyopic eye at randomization [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction (if applicable) by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  Best amblyopic eye visual acuity was computed as the better of the initial test and retest visual acuities at randomization.
  logMAR | 0.43 (0.15) | 0.45 (0.16) | 0.44 (0.16)
Best distance visual acuity in the fellow eye at randomization [Number; unit: participants] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction (if applicable) by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  Best fellow eye visual acuity was computed as the better of the initial test and retest visual acuities at randomization.
  participants
    20/32 | 5 | 5 | 10
    20/25 | 17 | 21 | 38
    20/20 | 27 | 26 | 53
    20/16 | 34 | 34 | 68
Best distance visual acuity in the fellow eye at randomization [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction (if applicable) by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  Best fellow eye visual acuity was computed as the better of the initial test and retest visual acuities at randomization.
  logMAR | -0.01 (0.09) | 0.00 (0.09) | -0.01 (0.09)
Best interocular eye visual acuity difference at randomization [Mean (Standard Deviation); unit: logMAR lines] — Best interocular eye visual acuity difference was computed as difference between the best amblyopic eye visual acuity and the best fellow eye visual acuity at randomization.
  logMAR lines | 4.4 (1.6) | 4.5 (1.7) | 4.5 (1.7)
Refractive error in amblyopic eye at enrollment [Number; unit: participants]
  0 to <+1.00D | 9 | 3 | 12
  +1.00 D to <+2.00 D | 5 | 3 | 8
  +2.00 D to <+3.00 D | 2 | 4 | 6
  +3.00 D to <+4.00 D | 13 | 6 | 19
  +4.00 D or more | 54 | 70 | 124
Refractive error in amblyopic eye at enrollment [Mean (Standard Deviation); unit: Diopters] | 4.58 (2.26) | 5.27 (1.94) | 4.93 (2.12)
Refractive error in fellow eye at enrollment [Number; unit: participants]
  <0 D | 1 | 1 | 2
  0 to <+1.00D | 22 | 14 | 36
  +1.00 D to <+2.00 D | 30 | 19 | 49
  +2.00 D to <+3.00 D | 10 | 14 | 24
  +3.00 D to <+4.00 D | 4 | 12 | 16
  +4.00 D or more | 16 | 26 | 42
Refractive error in fellow eye at enrollment [Mean (Standard Deviation); unit: Diopters] | 2.10 (1.86) | 2.89 (2.06) | 2.50 (2.00)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of 10-week Amblyopic Eye Visual Acuity
Description: The masked 10-week amblyopic eye visual acuity scores were tabulated for both treatment groups, and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The primary outcome analysis followed the intent-to-treat principle and included data from 10-week visual acuity exams completed between 8 and 15 weeks (inclusive) with no imputation for missing data.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
participants
  20/200 | 1 | 0
  20/160 | 0 | 0
  20/125 | 3 | 3
  20/100 | 3 | 2
  20/80 | 8 | 4
  20/63 | 6 | 9
  20/50 | 19 | 15
  20/40 | 23 | 20
  20/32 | 14 | 15
  20/25 | 3 | 12
  20/20 | 2 | 2
  20/16 | 0 | 0

2. Secondary Outcome: Compliance With Prescribed Patching by Treatment Group at 10 Weeks
Description: The distribution of compliance with prescribed treatment was tabulated for the 10-week outcome and as averaged scores across all study follow-up visits. Compliance was evaluated as excellent (>75%), good (51%-75%), fair (26%-50%), or poor (<26%) based on discussions with the parent and by reviewing study calendars maintained by the parent, who recorded the number of hours the child patched each day.
Time Frame: 10 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  Excellent | 66 | 59
  Good | 10 | 14
  Fair | 0 | 5
  Poor | 2 | 4
  Missing (Not applicable) | 4 | 1

3. Secondary Outcome: Average Compliance With Prescribed Patching by Treatment Group
Description: as for outcome 2
Time Frame: 10 weeks after randomization or later
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  Excellent | 65 | 60
  Good | 11 | 15
  Fair | 1 | 4
  Poor | 2 | 4
  Missing (Not applicable) | 3 | 0
  Treatment not per protocol | 0 | 1

4. Secondary Outcome: Treatment Group Comparison of the Proportion of Participants Who Have Improved by 2 or More logMAR Visual Acuity Lines at 10 Weeks Since Randomization
Description: The proportion of participants who improved at least 2 logMAR lines since randomization was computed at the 10-week outcome.
  The secondary outcome analysis was a treatment group comparison of the proportion of participants whose 10-week masked amblyopic eye visual acuity improved at least 2 logMAR lines since randomization using logistic regression, adjusting for visual acuity at randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
participants | 15 | 33
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Test type: Superiority or Other; p = 0.003, Regression, Logistic; The logistic regression model included amblyopic eye visual acuity at randomization as an adjustment covariate; Risk difference (unadjusted) = 22, 95% CI 2-sided [8 to 35]

5. Secondary Outcome: Treatment Group Comparison of 10-week Interocular Difference
Description: The secondary outcome analysis was a treatment group comparison of the 10-week interocular difference (IOD), computed as the difference between the masked amblyopic and fellow eye visual acuities, using an analysis of covariance (ANCOVA) model, adjusting for IOD at randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
logMAR lines | 3.7 (2.2) | 3.2 (2.1)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Test type: Superiority or Other; p = 0.01, ANCOVA; The ANCOVA model included interocular difference at randomization as an adjustment covariate; Mean Difference (Net) = 0.5, 95% CI 2-sided [0.1 to 1.0]

6. Secondary Outcome: Distribution of Baseline Characteristics at the 10-week Outcome
Description: The number of participants was tabulated by treatment group within categorical levels of prespecified baseline subgroup factors for participants with 10-week visual acuity exams completed between 8 to 15 weeks (inclusive)according to principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included participants who completed 10-week exams between 8 and 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
participants
  Gender: Female | 43 (0.17) | 41 (0.16)
  Gender: Male | 39 (0.13) | 41 (0.14)
  Race/Ethnicity: White (non-Hispanic) | 56 (0.16) | 63 (0.14)
  Race/Ethnicity: Non-White/Hispanic | 26 (0.14) | 19 (0.17)
  Age at randomization: 3 to <5 years | 20 (0.17) | 23 (0.15)
  Age at randomization: 5 years or older | 62 (0.11) | 59
  Amblyopic eye VA at randomization: 20/80 or worse | 12 | 15
  Amblyopic eye VA at randomization: 20/63 | 17 | 21
  Amblyopic eye VA at randomization: 20/50 | 26 | 24
  Amblyopic eye VA at randomization: 20/40 or better | 27 | 22
  Cause of amblyopia: Strabismus | 16 | 15
  Cause of amblyopia: Anisometropia | 40 | 31
  Cause of amblyopia: Combined mechanism | 26 | 36

7. Primary Outcome: Mean 10-week Amblyopic Eye Visual Acuity
Description: The primary outcome analysis was a treatment group comparison of the masked 10-week amblyopic eye visual acuity using an analysis of covariance (ANCOVA) model, adjusting for visual acuity at randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
logMAR | 0.38 (0.19) | 0.33 (0.18)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; The primary analysis was a treatment group comparison of the masked 10-week amblyopic eye visual acuity using an analysis of covariance (ANCOVA) model, adjusting for visual acuity at randomization. The analysis was a 2-sided test for efficacy to test the null hypothesis of no treatment difference, assuming 90% power and a type I error rate of 5%; Test type: Superiority or Other; p = 0.002, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate; Mean Difference (Net) = 0.6, 95% CI 2-sided [0.3 to 1.0]

8. Primary Outcome: Distribution of the Change in Amblyopic Eye Visual Acuity at 10 Weeks From Randomization
Description: The change in 10-week amblyopic eye visual acuity scores since randomization was tabulated for both treatment groups, and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: Randomization to 10 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
participants
  3 or more logMAR lines worse | 1 | 0
  2 logMAR lines worse | 3 | 2
  1 logMAR line worse | 13 | 7
  No change (0 logMAR line) | 19 | 17
  1 logMAR line improved | 31 | 23
  2 logMAR lines improved | 13 | 19
  3 or more logMAR lines improved | 2 | 14

9. Primary Outcome: Mean Change in Amblyopic Eye Visual Acuity at 10 Weeks From Randomization
Description: The change in 10-week amblyopic eye visual acuity was computed for both treatment groups and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: Randomization to 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
logMAR lines | 0.5 (1.2) | 1.2 (1.4)

10. Secondary Outcome: Mean Amblyopic Eye Visual at Randomization According to Baseline Characteristics for 10-week Outcome
Description: Mean amblyopic eye visual acuity at randomization was computed by treatment group within categorical levels of prespecified baseline subgroup factors. The analysis included data from participants with 10-week exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included participants who completed 10-week exams between 8 and 15 weeks (inclusive) according to the principles of the primary outcome analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
logMAR
  Gender: Female | 0.44 (0.17) | 0.45 (0.16)
  Gender: Male | 0.41 (0.13) | 0.44 (0.14)
  Race/Ethnicity: White (non-Hispanic) | 0.42 (0.16) | 0.45 (0.14)
  Race/Ethnicity: Non-White/Hispanic | 0.43 (0.14) | 0.43 (0.17)
  Age at randomization: 3 to <5 years | 0.45 (0.14) | 0.44 (0.12)
  Age at randomization: 5 years or older | 0.42 (0.16) | 0.45 (0.16)
  Cause of amblyopia: Strabismus | 0.46 (0.17) | 0.43 (0.15)
  Cause of amblyopia: Anisometropia | 0.39 (0.11) | 0.43 (0.13)
  Cause of amblyopia: Combined mechanism | 0.47 (0.19) | 0.46 (0.16)

11. Secondary Outcome: Treatment Comparison of Mean Amblyopic Eye Visual Acuity Change at 10-weeks According to Baseline Characteristics
Description: A treatment comparison of mean amblyopic eye visual acuity change since randomization was performed at the 10-week outcome according to categorical levels of prespecified baseline subgroup factors. The analysis included data from participants with 10-week exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 82
units on a scale
  Gender: Female | 0.4 (1.3) | 1.4 (1.3)
  Gender: Male | 0.7 (1.1) | 0.9 (1.5)
  Race/Ethnicity: White (non-Hispanic) | 0.5 (1.0) | 1.2 (1.4)
  Race/Ethnicity: Non-White/Hispanic | 0.5 (1.6) | 1.1 (1.3)
  Age at randomization: 3 to <5 years | 0.9 (1.0) | 1.5 (1.4)
  Age at randomization: 5 years or older | 0.4 (1.2) | 1.0 (1.4)
  Amblyopic eye VA at randomization: 20/80 or worse | 0.7 (1.4) | 1.3 (1.6)
  Amblyopic eye VA at randomization: 20/63 | 0.7 (1.3) | 1.6 (1.4)
  Amblyopic eye VA at randomization: 20/50 | 0.4 (1.2) | 1.4 (1.1)
  Amblyopic eye VA at randomization: 20/40 or better | 0.4 (1.1) | 0.5 (1.3)
  Cause of amblyopia: Strabismus | 1.1 (1.2) | 1.4 (1.3)
  Cause of amblyopia: Anisometropia | 0.3 (1.2) | 1.3 (1.5)
  Cause of amblyopia: Combined mechanism | 0.5 (1.1) | 1.0 (1.4)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; The treatment effect within gender was assessed by including an interaction term between treatment group and gender in the ANCOVA model, adjusting for amblyopic eye visual acuity at randomization and main effects corresponding to the interaction term; Test type: Superiority or Other; p = 0.04, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate
Statistical Analysis 2: Comparison: Control vs Intensified Treatment; The treatment effect within race/ethnicity was assessed by including an interaction term between treatment group and race/ethnicity in the ANCOVA model, adjusting for amblyopic eye visual acuity at randomization and main effects corresponding to the interaction term; Test type: Superiority or Other; p = 0.89, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate
Statistical Analysis 3: Comparison: Control vs Intensified Treatment; The treatment effect within age at randomization was assessed by including an interaction term between treatment group and age in the ANCOVA model, adjusting for amblyopic eye visual acuity at randomization and main effects corresponding to the interaction term; Test type: Superiority or Other; p = 0.49, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate
Statistical Analysis 4: Comparison: Control vs Intensified Treatment; The treatment effect within amblyopic eye visual acuity at randomization was assessed by including an interaction term between treatment group and visual acuity in the ANCOVA model, adjusting for the main effects corresponding to the interaction term; Test type: Superiority or Other; p = 0.37, ANCOVA
Statistical Analysis 5: Comparison: Control vs Intensified Treatment; The treatment effect within cause of amblyopia was assessed by including an interaction term between treatment group and amblyopia cause in the ANCOVA model, adjusting for amblyopic eye visual acuity at randomization and main effects corresponding to the interaction term; Test type: Superiority or Other; p = 0.50, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate

12. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity at Visit of Best Post-randomization Visual Acuity
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The distribution of best post-randomization (10 weeks or later) visual acuity scores in the amblyopic eye was tabulated for both treatment groups using the initial visual acuity score (if a retest was obtained.)
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  20/200 | 1 | 0
  20/160 | 0 | 0
  20/125 | 2 | 2
  20/100 | 3 | 3
  20/80 | 7 | 4
  20/63 | 7 | 7
  20/50 | 15 | 11
  20/40 | 16 | 21
  20/32 | 15 | 14
  20/25 | 12 | 15
  20/20 | 3 | 5
  20/16 | 1 | 1

13. Secondary Outcome: Mean Amblyopic Eye Visual Acuity at Visit of Best Post-randomization Visual Acuity
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. A treatment comparison of mean amblyopic eye visual acuity at the visit of best post-randomization visual acuity (10 weeks or later) was performed using an analysis of covariance, adjusting for amblyopic eye visual acuity at randomization.
Time Frame: 10 weeks after randomization or later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR | 0.33 (0.21) | 0.30 (0.19)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Test type: Superiority or Other; ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate; Mean Difference (Net) = 0.5, 95% CI 2-sided [0.04 to 1.0]

14. Secondary Outcome: Distribution of the Change in Best Post-randomization Visual Acuity in the Amblyopic Eye
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The distribution of change in best post-randomization (10 weeks or later) visual acuity in the amblyopic eye since randomization was tabulated for both treatment groups using the initial visual acuity score (if a retest was obtained.)
Time Frame: Randomization to 10 weeks or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  3 or more logMAR lines worse | 1 | 0
  2 logMAR lines worse | 3 | 2
  1 logMAR line worse | 12 | 6
  No change (0 logMAR line) | 13 | 17
  1 logMAR line improved | 21 | 16
  2 logMAR lines improved | 22 | 21
  3 or more logMAR lines improved | 10 | 21

15. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity Since Randomization at Visit of Best Post-randomization Visual Acuity
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The mean change in amblyopic eye visual acuity since randomization was computed for both treatment groups based on the visit of best post-randomization visual acuity (10 weeks or later) using the initial visual acuity score (if a retest was obtained.)
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR lines | 0.9 (1.5) | 1.5 (1.6)

16. Secondary Outcome: Treatment Group Comparison of the Proportion of Participants Who Have Improved by 2 or More logMAR Visual Acuity Lines Based on Visual Acuity at Best Post-randomization Visit
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The proportion of participants who improved at least 2 logMAR lines since randomization was computed based on the best post-randomization visual acuity in the amblyopic eye. The initial visual acuity score was used if a retest was obtained.
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants | 32 | 42

17. Secondary Outcome: Distribution of Best Fellow Eye Visual Acuity at 10-week Outcome
Time Frame: 10 weeks after randomization
Population: The analysis includes data from participants who completed a 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  20/63 | 0 | 0
  20/50 | 1 | 0
  20/40 | 1 | 0
  20/32 | 5 | 8
  20/25 | 19 | 14
  20/20 | 20 | 31
  20/16 | 36 | 30

18. Secondary Outcome: Mean Best Fellow Eye Visual Acuity at 10-week Outcome
Time Frame: 10 weeks after randomization
Population: The analysis includes data from participants who completed a 10-week exam.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR | 0.00 (0.11) | 0.00 (0.10)

19. Secondary Outcome: Distribution of Best Fellow Eye Visual Acuity at Final Visit
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  20/63 | 1 | 0
  20/50 | 1 | 0
  20/40 | 1 | 0
  20/32 | 4 | 5
  20/25 | 15 | 18
  20/20 | 20 | 28
  20/16 | 40 | 32

20. Secondary Outcome: Mean Best Fellow Eye Visual Acuity at Final Visit
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR | -0.01 (0.12) | 0.00 (0.09)

21. Secondary Outcome: Distribution of Change in Best Fellow Eye Visual Acuity Since Randomization at 10 Weeks
Time Frame: 10 weeks after randomization
Population: The analysis includes data from participants who completed a 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  3 or more logMAR lines worse | 1 | 1
  2 logMAR lines worse | 0 | 0
  1 logMAR line worse | 14 | 16
  No change (0 logMAR line) | 58 | 49
  1 logMAR line improved | 8 | 17
  2 logMAR lines improved | 1 | 0
  3 or more logMAR lines improved | 0 | 0
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Fisher's exact test was used to compare the proportion of participants in each treatment group with a loss of 2 or more lines in the better of the initial test and retest (if indicated) fellow eye visual acuities at the 10-week exam; Test type: Superiority or Other; p > 0.99, Fisher Exact

22. Secondary Outcome: Mean Change in Best Fellow Eye Visual Acuity Since Randomization at 10 Weeks
Time Frame: 10 weeks after randomization
Population: The analysis includes data from participants who completed a 10-week exam.
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR lines | -0.10 (0.7) | -0.02 (0.7)

23. Secondary Outcome: Distribution of Change in Best Fellow Eye Visual Acuity Since Randomization at Final Visit
Time Frame: 10 weeks after randomization or later
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  3 or more logMAR lines worse | 2 | 0
  2 logMAR lines worse | 1 | 0
  1 logMAR line worse | 11 | 16
  No change (0 logMAR line) | 53 | 50
  1 logMAR line improved | 13 | 16
  2 logMAR lines improved | 2 | 1
  3 or more logMAR lines improved | 0 | 0
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Fisher's exact test was used to compare the proportion of participants in each treatment group with a loss of 2 or more lines in the better of the initial test and retest (if indicated) fellow eye visual acuities at the final exam; Test type: Superiority or Other; p = 0.12, Fisher Exact

24. Secondary Outcome: Mean Change in Best Fellow Eye Visual Acuity Since Randomization at Final Visit
Time Frame: 10 weeks after randomization or later
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
logMAR lines | -0.04 (0.9) | 0.02 (0.7)

25. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Scores at Randomization
Description: The Preschool Randot test measures random dot stereoacuity from 800 to 40 arc seconds (800, 400, 200, 100, 60, 40). Lower scores indicate better stereoacuity and subjects who fail the first level (800 seconds of arc) are assigned a score of >800.
  We administer a pretest, and those with a failed or uninterpretable score do not proceed with the Randot testing.
  The Preschool Randot test consists of 3 booklets each with 2 sets of 4 random dot shapes (one is blank, 3 are actual figures), which can be matched to non-stereo shapes on the opposite side of the booklets. There are six levels (seconds of arc) in the test with two levels in each book. Each level has 4 rectangles that contain 3 shapes and one blank.
Time Frame: Randomization
Population: The analysis includes all participants who completed the 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  Failed pretest | 10 | 7
  > 800 seconds of arc | 39 | 47
  800 seconds of arc | 10 | 8
  400 seconds of arc | 6 | 5
  200 seconds of arc | 4 | 7
  100 seconds of arc | 7 | 1
  60 seconds of arc | 2 | 0
  40 seconds of arc | 2 | 2
  Not done | 2 | 6

26. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Scores at 10 Weeks
Time Frame: 10 weeks after randomization
Population: The analysis includes all participants who completed the 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 82 | 83
participants
  Failed pretest | 8 | 7
  > 800 seconds of arc | 33 | 44
  800 seconds of arc | 13 | 10
  400 seconds of arc | 10 | 12
  200 seconds of arc | 5 | 6
  100 seconds of arc | 11 | 0
  60 seconds of arc | 0 | 2
  40 seconds of arc | 2 | 1
  Not done | 0 | 1

27. Secondary Outcome: Change in Randot Preschool Stereoacuity Level at 10-week Outcome Since Randomization
Time Frame: 10 weeks after randomization
Population: Change in stereoacuity level at 10 weeks was computed for participants with measureable stereoacuity at randomization and at the 10-week primary outcome exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 69 | 68
participants
  2 or more levels worse | 2 | 2
  Within 1 level | 62 | 59
  2 or more levels improved | 5 | 7
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; An Exact Wilcoxon rank sum test was used for the difference between treatment groups in the distribution of levels of change in Randot Preschool Stereoacuity from randomization to 10 weeks; Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Scores at Randomization for Participants With Anisometropic Amblyopia
Time Frame: Randomization
Population: The analysis includes participants with anisometropic amblyopia (no strabismus) who completed the 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 32
participants
  Failed pretest | 3 | 3
  > 800 seconds of arc | 15 | 17
  800 seconds of arc | 7 | 3
  400 seconds of arc | 5 | 2
  200 seconds of arc | 3 | 3
  100 seconds of arc | 3 | 1
  60 seconds of arc | 2 | 0
  40 seconds of arc | 1 | 2
  Not done | 1 | 1

29. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Scores at 10 Weeks for Participants With Anisometropic Amblyopia
Time Frame: 10 weeks after randomization
Population: The analysis includes participants with anisometropic amblyopia (no strabismus) who completed the 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 32
participants
  Failed pretest | 3 | 2
  > 800 seconds of arc | 11 | 17
  800 seconds of arc | 7 | 4
  400 seconds of arc | 6 | 4
  200 seconds of arc | 4 | 3
  100 seconds of arc | 7 | 0
  60 seconds of arc | 0 | 1
  40 seconds of arc | 2 | 1
  Not done | 0 | 0

30. Secondary Outcome: Change in Randot Preschool Stereoacuity Level at 10-week Outcome Since Randomization for Participants With Anisometropic Amblyopia
Time Frame: 10 weeks after randomization
Population: Change in stereoacuity level at 10 weeks was computed for participants with anisometropic amblyopia (no strabismus) who had measureable stereoacuity at randomization and at the 10-week primary outcome exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 35 | 28
participants
  2 or more levels worse | 0 | 2
  Within 1 level | 32 | 22
  2 or more levels improved | 3 | 4
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Control | Intensified Treatment
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/86
Other Adverse Events (participants affected / at risk) | 6/83 | 4/86
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=83) | Intensified Treatment (N=86)
New ocular deviation or worsening of preexisting deviation by at least 10 pd (Eye disorders) | 6 (7) | 4 (7)

LIMITATIONS AND CAVEATS:
A potential study limitation is that compliance with patching was based on discussions with the parent and by reviewing study calendars maintained by the parent, which not an objective measure of compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No